CLINICAL TRIAL: NCT00000844
Title: A Multicenter, Prospective, Randomized, Double-Blind, Placebo-Controlled Trial of Three Preparations of Low-Dose Oral Alpha Interferon in HIV-Infected Patients With CD4+ Counts >= 50 and <= 350 Cells/mm3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: DATRI 022; 11727 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Adjuvants, Immunologic; Administration, Oral; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Interferon-alpha
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Interferon Alfa-n3; interferon alfa-n1

INTERVENTIONS:
Drug: Interferon alfa-n3
Drug: Interferon alfa-n1

SUMMARY:
To evaluate the effects of three preparations of low-dose oral interferon alpha (i.e., Alferon LDO, Veldona, and Ferimmune) on HIV symptoms in HIV-infected patients. To evaluate differences in response to oral interferon alpha according to gender, race/ethnicity, and use of antiretrovirals.

Previous or ongoing clinical trials to test the efficacy of low-dose oral interferon alpha have produced different results, and it is not clear whether the differences were due to the interferon alpha products used or to problems in the study design. Therefore, three preparations will be compared to evaluate their potential efficacies.

DETAILED DESCRIPTION:
Previous or ongoing clinical trials to test the efficacy of low-dose oral interferon alpha have produced different results, and it is not clear whether the differences were due to the interferon alpha products used or to problems in the study design. Therefore, three preparations will be compared to evaluate their potential efficacies.

Patients are randomized to receive 6 months of Alferon LDO alone, Alferon with Veldona, Alferon with Ferimmune, or three placebos, with follow-up visits monthly.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Symptomatic HIV infection.
* CD4 count 50 - 350 cells/mm3.

Prior Medication:

Allowed:

* Prior antiretrovirals (dose must be stable for at least 6 weeks prior to study entry).
* Maintenance therapy for a chronic condition.

Exclusion Criteria

Patients with the following prior condition are excluded:

* Change in antiretroviral therapy within past 6 weeks.

Prior Medication:

Excluded:

* Oral IFN-alpha or other immune-based therapy within the past month.
* Therapy for any acute disease within the past week.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 560
Dates: Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alston B, Study Chair; Standiford H, Study Chair; Kumi J, Study Chair; Greaves W, Study Chair
Locations (15):
- United States (15):
  - King - Drew Med Ctr, Los Angeles, California
  - AIDS Community Research Consortium, Redwood City, California
  - Yale Univ / New Haven, New Haven, Connecticut
  - Med Ctr of Delaware / Wilmington Hosp, Wilmington, Delaware
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Abundant Life Clinic Foundation, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Henry Ford Hosp, Detroit, Michigan
  - Univ of Minnesota Hosp, Minneapolis, Minnesota
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Dr Barbara Justice, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - New York Med College / Westchester County Med Ctr, Valhalla, New York
  - Univ of Pennsylvania Med Ctr, Philadelphia, Pennsylvania
  - Meharry Med College, Nashville, Tennessee

REFERENCES:
- [Background] Randall P. Low-dose oral alpha interferon study opens. NIAID AIDS Agenda. 1996 Jun:4-5. PMID 11363808
- [Background] Low-dose oral alpha interferon trial closes. NIAID AIDS Agenda. 1997 Aug:10. PMID 11364607
- [Result] Alston B, Ellenberg JH, Standiford HC, Muth K, Martinez A, Greaves W, Kumi J. A multicenter, randomized, controlled trial of three preparations of low-dose oral alpha-interferon in HIV-infected patients with CD4+ counts between 50 and 350 cells/mm(3). Division of AIDS Treatment Research Initiative (DATRI) 022 Study Group. J Acquir Immune Defic Syndr. 1999 Dec 1;22(4):348-57. doi: 10.1097/00126334-199912010-00005. PMID 10634196